CLINICAL TRIAL: NCT00290472
Title: A Phase II Study of CCI-779 in B-cell Lymphoma and CLL
Brief Title: CCI-779 in Treating Patients With Recurrent or Refractory B-Cell Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00047; NCI-2009-00047 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000365314; NCI-6199; 12983A; 6199 (Other: University of Chicago); 6199 (Other: CTEP); N01CM62201 (NIH); N01CM62202 (NIH); P30CA014599 (NIH); NCT00084474 (obsolete NCT alias)
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2013-02

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Malignant Neoplasm; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Waldenstrom Macroglobulinemia | interventions — temsirolimus; Sirolimus

ARMS (1):
- Arm I (Experimental): Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 8 weeks.
  Interventions: Drug: temsirolimus

INTERVENTIONS:
Drug: temsirolimus
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel

SUMMARY:
Drugs used in chemotherapy, such as CCI-779, work in different ways to stop cancer cells from dividing so they stop growing or die. This phase II trial is studying how well CCI-779 works in treating patients with recurrent or refractory B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the complete and partial response rate in patients with recurrent or refractory B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia treated with CCI-779.

II. Determine the toxicity and safety of this drug in these patients. III. Correlate the degree of activation of P13/AKT/mTOR pathway and levels of CDK inhibitors with response in patients treated with this drug.

IV. Correlate CCI-779 induced inactivation of mTOR with response in these patients.

OUTLINE: Patients are stratified according to disease (aggressive lymphoma [group A] vs follicular lymphoma [group B] vs small lymphocytic lymphoma or chronic lymphocytic leukemia [group C]).

Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed B-cell non-Hodgkin's lymphoma, including the following subtypes:

  * Aggressive B-cell lymphoma (Group A)

    * Diffuse large B-cell lymphoma
    * Transformed lymphoma
  * Follicular lymphoma (Group B)
  * Small lymphocytic lymphoma

    * Chronic lymphocytic leukemia (CLL) (Group C)
    * Other B-cell small lymphocytic disorders
* No mantle cell lymphoma
* No potentially curative treatment options because of lack of response, relapse, or ineligibility
* Relapsed or refractory disease
* Patients with refractory disease (i.e., less than a partial response to the last treatment) must have received no more than 3 prior regimens (group A)
* Patients with sensitive disease (i.e., at least a partial response to the last treatment) must have received no more than 4 prior regimens (group A)
* Patients who have failed prior autologous transplantation are eligible (group A)

  * No more than 5 prior regimens (groups B and C)
  * The salvage regimen, conditioning regimen, and any maintenance therapy are considered 1 regimen
* Prior rituximab or alemtuzumab is not considered prior therapy
* No limitation to the amount of prior radiotherapy
* No CNS involvement
* Performance status: ECOG 0-2 OR Karnofsky 60-100%
* Life expectancy more than 3 months
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to CCI-779
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other active malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix Completed therapy and considered < 30% risk of relapse
* No other concurrent uncontrolled illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent prophylactic hematopoietic colony-stimulating factors
* No concurrent pegfilgrastim
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* More than 4 weeks since prior radiotherapy and recovered
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent unconventional therapies, food, or vitamin supplements containing Hypericum perforatum (St. John's wort)
* No other concurrent known inducers of CYP3A4
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* Measurable disease*

  * At least 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan [Note: *Only bone marrow or peripheral blood involvement required for CLL and Waldenstrom's macroglobulinemia ]
* Absolute neutrophil count >= 1,000/mm3
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* AST and ALT =< 2.5 times ULN
* Creatinine =< 1.5 times ULN
* Fasting cholesterol =< 350 mg/dL
* Fasting triglycerides =< 400 mg/dL
* Platelet count >= 50, 000/mm3 (> 20,000/mm3 for patients with thrombocytopenia due to bone marrow involvement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2004-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Smith, Principal Investigator — University of Chicago
Locations (13):
- United States (13):
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Evanston Hospital CCOP, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Adventist La Grange Memorial Hospital, La Grange, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Iowa, Iowa City, Iowa
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - M D Anderson Cancer Center, Houston, Texas
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Smith SM, van Besien K, Karrison T, Dancey J, McLaughlin P, Younes A, Smith S, Stiff P, Lester E, Modi S, Doyle LA, Vokes EE, Pro B. Temsirolimus has activity in non-mantle cell non-Hodgkin's lymphoma subtypes: The University of Chicago phase II consortium. J Clin Oncol. 2010 Nov 1;28(31):4740-6. doi: 10.1200/JCO.2010.29.2813. Epub 2010 Sep 13. PMID 20837940

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient never received protocol treatment and was excluded from analysis.
Groups:
- Aggressive B-cell Lymphoma: Patients received Temsirolimus (CCI-779) IV over 30 minutes on days 1,8,15, and 22. Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients were followed every 8 weeks. Aggressive B-cell lymphoma group was defined as patients with histologic subtypes included diffuse large B-cell lymphoma and transformed follicular lymphoma.
- Follicular Lymphoma: Patients received Temsirolimus (CCI-779) IV over 30 minutes on days 1,8,15, and 22. Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients were followed every 8 weeks. Follicular lymphoma group was defined as patients with histologic subtypes included follicular lymphoma.
- Chronic Lymphocytic Leukemia: Patients received Temsirolimus (CCI-779) IV over 30 minutes on days 1,8,15, and 22. Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients were followed every 8 weeks. Chronic lymphocytic leukemia group was defined as patients with histologic subtypes included chronic lymphocytic leukemia, small lymphocytic lymphoma, and other indolent lymphomas.
Period: Overall Study
Arm/Group | Aggressive B-cell Lymphoma | Follicular Lymphoma | Chronic Lymphocytic Leukemia
Started | 32 | 39 | 18
Completed | 32 | 39 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aggressive B-cell Lymphoma | Follicular Lymphoma | Chronic Lymphocytic Leukemia | Total
Number analyzed (Participants) | 32 | 39 | 18 | 89
Age, Continuous [Median (Full Range); unit: years] | 67 [30 to 87] | 59 [28 to 75] | 57 [38 to 82] | 61 [28 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 7 | 37
  Male | 17 | 24 | 11 | 52

OUTCOME MEASURES:

1. Primary Outcome: Objective Overall Response Rate
Description: The 1999 international response criteria (http://www.ncbi.nlm.nih.gov/pubmed/10655437#) as published by Cheson was used for the definition of target lesions and CT scans were used for response assessment. CR(complete response)/CRu(unconfirmed complete response) requires disappearance of all target lesions; PR (partial response) requires >=50% decrease in the sum of the products of the greatest diameters; Overall Response (OR)=CR/CRu+PR.
Time Frame: Up to 6 years
Measure: Number; unit: percentage of participants
Arm/Group | Aggressive B-cell Lymphoma | Follicular Lymphoma | Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 32 | 39 | 18
percentage of participants | 28.1 | 53.8 | 11.1

2. Primary Outcome: Duration of Response
Description: Duration of response was the time from date of response to date of progression and evaluated among participants with response. According to the 1999 international response criteria as published by Cheson, progression/progressive disease is defined as >=50% increase from nadir in the sum of the products of the greatest diameters of any previously identified abnormal node for PRs or nonresponders, or appearance of any new lesion during or at the end of therapy.
Time Frame: Up to 6 years
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Aggressive B-cell Lymphoma | Follicular Lymphoma | Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 9 | 21 | 2
Month | 2.4 [2.1 to 28.4] | 13.3 [6.2 to 16.5] | NA [NA to NA] — Chronic Lymphocytic Leukemia group had no progression events.

3. Primary Outcome: Overall Survival
Description: The overall survival was evaluated using the Kaplan-Meier estimator.
Time Frame: Up to 6 years
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Aggressive B-cell Lymphoma | Follicular Lymphoma | Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 32 | 39 | 18
Month | 7.3 [4.3 to 18.1] | NA [NA to NA] — The median Overall Survival and the associated 95% CI was not reached. | 31.5 [9.5 to NA] — The upper limit of the 95% CI interval was undetermined due to the heavy censoring.

ADVERSE EVENTS:
Groups:
- Temsirolimus: All patients
Arm/Group | Temsirolimus
Serious Adverse Events (participants affected / at risk) | 21/89
Other Adverse Events (participants affected / at risk) | 89/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus (N=89)
Anorectal infection (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dysphagia, esophagitis, odynophagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Hemorrhage (Gastrointestinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia (Infections and infestations) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Pyrexia (General disorders) | 1
Renal/Genitourinary-other (Renal and urinary disorders) | 1
Respiratory tract infection NOS (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Stomatitis/pharyngitis (Gastrointestinal disorders) | 1
Thrombosis/ embolism (Vascular disorders) | 1
Tooth infection (Infections and infestations) | 1
Urinary retention (Renal and urinary disorders) | 1
Vulvitis (Infections and infestations) | 1
Oseophagitis NOS (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus (N=89)
Abdominal pain (Gastrointestinal disorders) | 13
Alanine aminotransferase increased (Investigations) | 27
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 16
Anorexia (Metabolism and nutrition disorders) | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Aspartate aminotransferase increased (Investigations) | 34
Back pain (Musculoskeletal and connective tissue disorders) | 7
Blood alkaline phosphatase intreased (Investigations) | 23
Blood creatinine increased (Investigations) | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 11
CD4 lymphocytes decreased (Investigations) | 5
Chills (General disorders) | 5
Constipation (Gastrointestinal disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 31
Death (General disorders) | 22
Diarrhea (Gastrointestinal disorders) | 24
Disease progression (General disorders) | 8
Dizziness (Nervous system disorders) | 10
Dry mouth (Gastrointestinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20
Ear, nose and throat examination abnormal (General disorders) | 25
Edema (General disorders) | 29
Edema : limb (General disorders) | 6
Eye disorder (Eye disorders) | 5
Eye problem (Eye disorders) | 6
Fatigue (General disorders) | 56
Fever (General disorders) | 15
General symptom (General disorders) | 5
Headache (Nervous system disorders) | 19
Hemoglobin (Blood and lymphatic system disorders) | 63
Hemorrhage nasal (Blood and lymphatic system disorders) | 8
Hypercholesterolemia (Metabolism and nutrition disorders) | 44
Hyperglycemia (Metabolism and nutrition disorders) | 50
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hypertriglyceridemia (Metabolism and nutrition disorders) | 59
Hypoalbuminemia (Metabolism and nutrition disorders) | 24
Hypocalcemia (Metabolism and nutrition disorders) | 20
Hypokalemia (Metabolism and nutrition disorders) | 25
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypophsphatemia (Metabolism and nutrition disorders) | 19
Hypotension (Vascular disorders) | 6
Infection (Infections and infestations) | 21
Insomnia (Psychiatric disorders) | 7
Leukopenia (Blood and lymphatic system disorders) | 65
Lymphopenia (Blood and lymphatic system disorders) | 42
Memory impairment (Nervous system disorders) | 5
Mood alteration-depression (Psychiatric disorders) | 6
Muscle weakness (Musculoskeletal and connective tissue disorders) | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Nausea (Gastrointestinal disorders) | 19
Neuropathy-sensory (Nervous system disorders) | 16
Neutrophil count (Investigations) | 52
Oral pain (Gastrointestinal disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Pain - other (General disorders) | 6
Platelet count decreased (Investigations) | 73
Proteinuria (Renal and urinary disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Pyrexia (General disorders) | 6
Rash desquamating (Skin and subcutaneous tissue disorders) | 25
Rash/dermatitis (Skin and subcutaneous tissue disorders) | 20
Stomatitis/ pharyngitis (Gastrointestinal disorders) | 29
Sweating (General disorders) | 6
Taste alteration (Gastrointestinal disorders) | 8
Upper respiratory infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 6
Vomiting (Gastrointestinal disorders) | 11
Pharyngolaryngea (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less